#### **Protocol title:**

# Infrared and Broadband Light for Skin Aging NCT03243981

Version date 06162016

Principal Investigator:

Anne Lynn S. Chang, MD
Assistant Professor of Dermatology
Stanford University School of Medicine
450 Broadway Street, MC 5334
Redwood City, CA 94305
Phone 650 644 7318
alschang@stanford.edu

Co-investigator:

Patrick Bitter, MD Tyler Hollmig, MD

Sponsor:

Sciton

## **Primary Objectives**

- -To assess the effect of broadband light with skin tightening properties on the gene expression pattern of aging skin
- -To assess the duration of the skin rejuvenation effects of broadband light with skin tightening properties (optional)

## Background

Studies in model organisms suggest that aged cells can be functionally rejuvenated, but whether this concept applies to human skin is unclear. Recently, we applied 3'-end sequencing for expression quantification ("3-seq") to discover the gene expression program associated with human photoaging and intrinsic skin aging (collectively termed "skin aging"), and the impact of broadband light (BBL) treatment. We found significant changes in 2,265 coding and noncoding RNAs, of which 1,293 that became "rejuvenated" after BBL treatment, whereby they became more similar to their expression level in youthful skin. Rejuvenated genes (RGs) included several known key regulators of organismal longevity and their proximal long noncoding RNAs. Hence, BBL treatment can restore gene expression pattern of photo-aged and intrinsically aged human skin to resemble young skin.

However, the duration of these effects and the potential to augment these effects through increases in particular wavelengths of light have not been explored. The Sciton SkinTyte (800-1800nm) is the ideal technology to examine these questions, since this device has been used in the clinical setting to reduce cheek and submental laxity (Gold, 2010). It incorporates the broadband light technology with an emphasis on 590 nm filter to achieve these clinical results.

## **Study Procedures**

The design of this study is a prospective, single blind study of six adult volunteers.

#### Human subjects and sample acquisition

This study will be conducted in accord with Declaration of Helsinki principles. After Institutional Review Board approval and informed consent is obtained, six female participants over the age of 55 years will undergo BBLST treatments to the left forearm. Inclusion criteria included Fitzpatrick skin type II or III, and a global assessment of forearm skin aging consistent with moderate or severe forearm skin aging (modified validated instrument from McKenzie *et al.*, 2011) for treated participants. Treatments will be performed on the Sciton Joule Platform using BBL in Skintyte mode with 590ST filter. On a separate part of the arm that is clearly marked, Skintyte alone will be applied. Untreated areas will also be marked. All markings will be photographed. The same investigator will perform the treatments at 4-week intervals for a total of 3 treatments. At each

treatment session, two or more passes were performed. Four weeks after the third BBL treatment, 4 mm skin biopsies will performed by Keys punch technique from the BBLST treated, ST treated and adjacent untreated skin. These specimens will be bisected and placed into either RNAlater (Ambion Cat# AM7022) or formalin solution for with H&E, von Giesen or PAS staining.

## Inclusion criteria

- 1. Female
- 2. Age 55 years or older (total 6)
- 3. Fitzpatrick skin type 2-3
- 4. Photo-aging at least moderate on the extensor forearms

## Exclusion criteria

- 1. Unable to understand and sign informed consent form
- 2. Unable to comply with study procedures
- 3. Pregnant or lactating
- 4. Prior treatment to forearms including topical retinoid, laser treatment, photodynamic treatment, prescription topical agents x 1 month
- 5. Active skin conditions that precluding treatment including zoster, blistering skin disease, psoriasis, atopic dermatitis, abnormal scarring, skin cancer in the area of study treatment
- 6. Currently on hormone based therapy (both systemic and topical)

#### Screening visit

After written informed consent signing, subjects will undergo the following procedures, eligibility will be assessed and the following will be obtained:

- Demographics
- Medical Histories
- Physical Examination
- Photographs with high resolution digital camera
- Cutometry

Baseline (visit 1, treatment #1), Day 28 visit (treatment #2), Day 56 visit (treatment #3)

Each subject would have three treatments at one month intervals by the same health care provider. Each subject would have three biopsies at approximately one month post treatment (day 84 visit). The biopsies will be of the BBL treated, the BBL-ST treated and the untreated. Total biopsy per patient at the end of the study is 3.



#### Clinical characteristics

Mean ages, skin type and medical histories will be described. The mean elasticity and transepidermal water loss will be described for treated (day 84 and possibly 168), untreated (day 84 or day 168 (if we go with the latter budget scenario)). The degree of fine wrinkling, sagging, texture, erythema and overall appearance will be assessed using a 5-point Likert scale and compared for treated, untreated and young skin. T-tests will be used to assess the mean, standard deviations and p values at a significance level <0.05 as described in Chang *et al.*, 2013.

#### 3-Seq and bioinformatics

Total RNA will be extracted using RNeasy Fibrous Tissue Mini Kit (Qiagen). 3-seq will be performed as described in Beck AH *et al.*, 2010. In brief, oligo-dT-directed reverse transcription generated cDNAs corresponding to 3' ends of poly-adenylated transcripts; the cDNAs were cloned and subjected to deep sequencing on the Illumina GAIIx platform with raw read length 36bp. Raw reads were aligned to human genome (hg18) using bowtie (Langmead *et al.*, 2009); each sample generated 6.5-12.4 million uniquely mappable reads. 3' sequencing of skin transcripts was performed to assess length distributions. Reads Per Kilobase of exon per Million mappable reads (RPKM, a direct measure of transcript abundance) and the number of raw reads falling on to each gene will be calculated using self-developed script by K. Qu. RefSeq (www.ncbi.nlm.nih.gov/RefSeq) and Ensembl (http://www.ensembl.org) annotated noncoding genes were included. Significant genes will be called using DESeq package (http://www.bioconductor.org) comparing aged-treated versus aged-untreated samples (genes changed due to treatment), and aged-untreated

versus young-untreated (genes changed due to aging). Unsupervised hierarchical clustering of significantly different expressed genes will be performed using Cluster. Treated versus untreated skin across the time points of Study Day 28 and Day 56 will analyzed. The young group will serve as the comparison group. 3'-seq technique will allow for analysis of long non-coding RNAs.

Gene Otology terms were generated using DAVID Bioinformatics Resources 6.7 (http://david.abcc.ncifcrf.gov/). Genes close to IncGenes will identified using GREAT database (http://great.stanford.edu). This data will be deposited into the Gene Expression Omnibus (GEO).

## RT-qPCR

Total RNA will be extracted with TRIzol (Invitrogen) followed by RNeasy column purification (Qiagen) and DNAse Turbo Treatment (Ambion). RT-qPCR was performed using total RNA (10 ng), Taqman One Step RT-PCR master mix, and one of the following Taqman assays: GAPDH (Hs99999905\_m1) and ZMPSTE24 (Hs00956778\_m1) (Applied Biosystems). Reactions will be in triplicate for each sample and performed a minimum of two times. Data will be normalized to GAPDH levels.

# Study Endpoints

-effect of broadband light with skin tightening properties on the gene expression pattern of aging skin as measured by 3'-end sequencing, between treated and untreated

-duration of the skin rejuvenation effects of broadband light with skin tightening properties including cutometry, transepidermal water loss, sagging, fine wrinkling, coarse wrinkling and physician global assessment between pre-treatment, day 84 (one month after last treatment) (and possibly day 156 (2 months after last treatment) if budget allows).

#### References

Adams S, Pankow S, Werner S, Munz B (2007). Regulation of NFKB activity and keratinocytic differentiation by the RIP4 protein: implications for cutaneous wound repair. *JID* 127(3): 538-44.

Adler AS, Sinha S, Kawahara TLA, et al. (2007). Motif module map reveals enforcement of aging by continual NFKB activity. Genes and Dev 21:3244-57.

Beck AH, Weng Z, Witten DM, et al. (2010). 3'-end sequencing for expression quantification (3SEQ) from archival tumor samples. PLoS One 19; 5(1): e8768.

Bernard D, Gosselin K, Monte D *et al.* (2004) Involvement of Rel/ NFkB transcription factors in keratinocyte senescence. *Cancer Res* 64: 472-81.

Caslini C, Connelly JA, Serna A, *et al.* (2009). MLL associates with telomeres and regulates telomeric repeat-containing RNA transcription. *Mol Cell Biol* 29 (No. 16): 4519-4526.

Chang A, Bitter PB *et al.* (2013) Rejuvenation of gene expression pattern of aged human skin by broadband light. J of Investig Dermatol 133(6): 1691.

Chang HY, Nuyten DS, Sneddon JB *et al.* (2005). Robustness, scalability and integration of a wound-response gene expression signature in predicting breast cancer survival. *PNAS USA* 102(10): 3738-3743.

Chen C, Liu Y, Liu Y, Zheng P. (2009) mTOR regulation and therapeutic rejuvenation of aging hematopoietic stem cells. *Sci Signal*. 2(98): p.ra71.

Curran SP, Ruvkun G (2007). Lifespan regulation by evolutionarily conserved genes essential for viability. *PLoS Genet* 3(4):e56.

ENCODE Consortium (2011). The user's guide to the encyclopedia of DNA elements. *PLoS Biology* 9(4): 1001046.

Fisher GJ, Varani J, Voorhees JJ (2008). Looking older: fibroblast collapse and therapeutic implications. Arch Dermatol 144 (5).

Gold MH (2010). Update on tissue tightening. *Journal of clinical and aesthetic dermatology*. 3(5).

Goldberg DJ (2000). New collagen formation after dermal remodeling with an intense pulsed light source. *J Cutan Laser Ther* 2:59-61.

Greer EL, Maures TJ, Hauswirth AG, *et al.* (2010). Members of the histone H3 lysine 4 trimethylation complex regulate lifespan in germline-dependent manner in c. elegans. *Nature* 466(7304):383-387.

Gupta RA, Shah N, Wang KC, *et al.* (2010). Long non-coding RNA HOTAIR reprograms chromatin state to promote cancer metastasis. *Nature* 464:1071-1076.

Holzenberger M, Dupont J, Ducos B *et al.* (2003). IGF1 receptor regulates lifespan and resistance to oxidative stress in mice. *Nature* 421:182-185.

Hsieh C-C, Kuro-o M, Rosenblatt KP, *et al.* (2010). The ASK1-Signalosome regulates p38 MAPK activity in response to levels of endogenous oxidative stress in the Klotho mouse models of aging. *Aging* 2(9):597-611.

Itahana K, Zou Y, Itahana Y, *et al.* (2003). Control of the replicative life span of human fibroblasts by p16 and the polycomb protein Bmi-1. *Mol Cell Biol* 23 (No. 1):389-401.

Kirby K, Hu J, Hilliker AJ, Phillips JP (2002). RNA interference-mediated silencing of Sod2 in Drosophila leads to early adult-onset mortality and elevated endogenous oxidative stress. *PNAS* 99(25): 16162-7.

Langmead B, Trapnell C, Pop M, *et al.* (2009). Ultrafast and memory-efficient alignment of short DNA sequences to the human genome. *Genome Biology* 10:R25

Lee Y, Kim H, Kim S *et al.* (2009). Activation of toll-like receptors 2, 3, or 5 induces matrix metalloproteinase-1 and -9 expression with the involvement of MAPKs and NFkB in human epidermal keratinocytes. *Experimental Dermatology*, 19: e44-49.

Liu L, Rando TA (2011). Manifestations and mechanisms of stem cell aging. *JCB* 103 (No. 2):257-266.

Loewer S, Cabili MN, Guttman M, *et al.* (2010). Large intergenic non-coding RNA-RoR modulates reprogramming of human induced pluripotent stem cells. *Nature Genetics* 42:1113-1117.

Long X, Spycher C, Han ZS, *et al.* (2002). TOR deficiency in C. elegans causes developmental arrest and intestinal atrophy by inhibition of mRNA translation. *Curr Biol* 12: 1448-61.

de Magalhaes JP, Wuttke D, Wood SH, *et al.* (2012). Genome-environment interactions that modulate aging: powerful targets for drug discovery. *Pharmacol Rev* 64(1):88-101.

Mayr C, Bartel DP (2009). Widespread shortening of 3'UTRs by alternative cleavage and polyadenylation activates oncogenes in cancer cells. *Cell* 138(4):673-84.

McKenzie NE, Saboda K, Duckett LD *et al.* (2010). Development of a photographic scale for consistency and guidance in dermatologic assessment of forearm sun damage. *Arch Dermatol* 147 (1): 31-36.

Mehler MF, Mattick JS (2007). Noncoding RNAs and RNA editing in brain development, functional diversification, and neurological disease. *Physiol Rev* 87 (No. 3):799-823.

Morozova O, Hirst M, and Marra MA (2009). Applications of new sequencing technologies for transcriptome analysis. *Annu Rev Genomics Hum Genet* 10:135-51.

Nelson TJ, Behfar A, Yamada S, et al. (2009). Stem cell platforms for regenerative medicine. Clinical and Translational Science 2(3):222-227.

Negishi K, Tezuka Y, Kushikata N, *et al.* (2001). Photorejuvenation for Asian Skin by Intense pulsed light. *Dermatol Surg* 27:627-31.

Paddock HN, Schultz GS, Baker HV *et al.* (2003). Analysis of gene expression patterns in human postburn hypertrophic scars, *J Burn Care Rehabil* 24(6): 371-7.

Parado J, Bougria M, Ayala A, *et al.* (1999). Effects of aging on the various steps of protein synthesis: fragmentation of elongation factor 2. *Free Radic Biol Med* 26:362-370.

Partridge L (2010). The new biology of ageing. *Phil Trans R Soc B 12* 365 (No. 1537): 147-154.

Prieto VG, Sadick NS, Lloreta J, *et al.* (2002). Effects of intense pulsed light on sun-damaged human skin, routine, and ultra-structural analysis. *Lasers Surg Med* 30:82-5.

Rodwell G, Sonu R, Zahn JM, *et al.* (2004). A transcriptional profile of aging in the human kidney. *PLoS Biology* 2(12).

Serrano M (2011). Cancer: final act of senescence. Nature 479, 481-482.

Shapiro, IM, Cheng, AW, Flytzanis, NC *et al.* (2011). An EMT-driven alternative splicing program occurs in human breast cancer and modulates cellular phenotype. *PLoS Genet.* 7, e1002218.

Shaw T, Martin P (2009) Epigenetic reprogramming during wound healing: loss of polycomb-mediated silencing may enable upregulation of repair genes. *EMBO reports* 10 (8): 881-6

Tariq M, Kim HJ, Jejelowo O, *et al.* (2011). Whole-transcriptome RNAseq analysis from minute amount of total RNA. *Nucl. Acids Res.* 

Wang Z, Gersten M, Snyder M (2009). RNA-Seq: a revolutionary tool for transcriptomics. *Nat Rev Genet* 10(1): 57-63.

Wapinski O, Chang HY (2011). Long noncoding RNAs and human disease. *Trends in Cell Biology* 21(6): 354-61.